CLINICAL TRIAL: NCT05006716
Title: A Phase 1/2, Open-Label, Dose-Escalation and -Expansion Study of the Bruton Tyrosine Kinase Targeted Protein Degrader BGB-16673 in Patients With B-Cell Malignancies
Brief Title: A Dose-Escalation and Expansion Study of BGB-16673 in Participants With B-Cell Malignancies
Acronym: CaDAnCe-101
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-16673-101; 2022-502157-33-00 (Other: EU CT Number)
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: B-cell Malignancy; Marginal Zone Lymphoma; Follicular Lymphoma; Non-Hodgkin Lymphoma; Waldenström Macroglobulinemia; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Mantle Cell Lymphoma; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Part 1a (Monotherapy Dose Escalation) (Experimental): Dose escalation in specific subtypes of non-Hodgkin lymphoma (NHL), including relapsed or refractory (R/R) marginal zone lymphoma (MZL), R/R follicular lymphoma (FL) Grades 1, 2, and 3a, R/R mantle cell lymphoma (MCL), R/R chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), R/R diffuse large B-cell lymphoma (DLBCL), R/R Richter's transformation (RT), and R/R Waldenström macroglobulinemia (WM), to evaluate the safety and tolerability of BGB-16673.
  Interventions: Drug: BGB-16673
- Part 1b (Monotherapy Safety Expansion) (Experimental): Participants with R/R MZL, MCL, CLL/SLL, and WM will be enrolled at selected doses to help determine the recommended dose(s) for expansion (RDFE(s)) for BGB-16673.
  Interventions: Drug: BGB-16673
- Part 1c (Additional Monotherapy Safety Expansion) (Experimental): Additional safety data will be collected from participants with R/R MZL, WM, RT, DLBCL, or FL to confirm the RDFE(s) of BGB-16673 for those with non-CLL/SLL/MCL histologies.
  Interventions: Drug: BGB-16673
- Part 1d (Additional Monotherapy Safety Expansion in R/R CLL/SLL) (Experimental): Participants with R/R CLL/SLL will be enrolled at selected RDFE(s) to generate additional safety and efficacy data for BGB-16673.
  Interventions: Drug: BGB-16673
- Part 1e (Japan-only Cohort) (Experimental): Japanese participants with R/R MZL, FL, MCL, CLL/SLL, and WM will be enrolled at selected RDFE(s) to assess the safety and tolerability of BGB-16673.
  Interventions: Drug: BGB-16673
- Part 1f (Additional Monotherapy Safety Expansion in BTKi Naive B-Cell Malignancies) (Experimental): Participants with CLL/SLL, MCL, WM, MZL, or Richter's transformation to DLBCL who have not received a prior BTKi (either covalent or noncovalent) will be enrolled at selected dose levels.
  Interventions: Drug: BGB-16673
- Phase 2 (Monotherapy Expansion) (Experimental): Cohorts of participants with R/R CLL/SLL, R/R MCL, R/R WM, R/R MZL, R/R FL, R/R RT, and R/R DLBCL will be enrolled to receive the RDFE(s) identified in Phase 1 to further evaluate the safety and efficacy of BGB-16673.
  Interventions: Drug: BGB-16673

INTERVENTIONS:
Drug: BGB-16673 — Orally administered

SUMMARY:
Study consists of two main parts to explore BGB-16673 recommended dosing, a Phase 1 monotherapy dose finding comprised of monotherapy dose escalation and monotherapy safety expansion of selected doses, and a Phase 2 (expansion cohorts)

DETAILED DESCRIPTION:
Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria :

1. Confirmed diagnosis (per World Health Organization (WHO) guidelines, unless otherwise noted) of one of the following: Marginal Zone Lymphoma (MZL), R/R follicular lymphoma (FL), mantle cell lymphoma (MCL), chronic lymphocytic leukemia and small lymphocytic lymphoma (CLL/SLL), Waldenström macroglobulinemia (WM), R/R diffuse large B-cell lymphoma (DLBCL), or Richter's transformation to DLBCL.
2. Participants who have previously received a covalently-binding Bruton´s tyrosine kinase (BTK) inhibitor (BTKi) in any line of therapy must have received treatment with the BTK inhibitor for ≥ 8 weeks (unless reason for discontinuation is intolerance).
3. For dose-finding and dose-expansion, participants who had previously received a covalently-binding BTK inhibitor as monotherapy or in combination with other anticancer agents are eligible for the study if they meet any of the following criteria: discontinued the previous BTK inhibitor due to disease progression, experienced disease progression after completing treatment with a BTK inhibitor or discontinued the BTK inhibitor due to toxicity or intolerance.
4. Measurable disease by radiographic assessment or serum IgM level (WM only)
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
6. Participants enrolling in the dose finding phase of the study may be previously treated with a BTKi or may be naïve to BTKi therapy depending on the diagnosis and country of enrollment; participants with MCL enrolling in the expansion cohorts (Phase 2) must have been treated with a BTKi in a prior line of therapy; CLL/SLL participants, in addition to being treated with a BTKi in a prior line of therapy, must also have received a Bcl-2 inhibitor in a prior line of therapy as well (Phase 2).

Exclusion Criteria:

1. Prior malignancy (other than the disease under study) within the past 2 years, except in situ malignancies that have been curatively resected, localized breast cancer treated with curative intent with no evidence of breast active disease for more than 3 years and receiving adjuvant hormonal therapy, localized Gleason score ≤ 6 prostate cancer undergoing observation or treatment with androgen depravation, or any other cancer treated with curative intent, not on adjuvant treatment, and in the opinion of the investigator is unlikely to recur.
2. Requires ongoing systemic treatment for any other malignancy
3. Requires ongoing systemic (defined as ≥ 10 mg/day of prednisone or equivalent) corticosteroid treatment.
4. Current or history of central nervous system involvement including the brain, spinal cord, leptomeninges, and cerebrospinal fluid (as documented by imaging, cytology, or biopsy) by B-cell malignancy, regardless of whether participants had received treatment for central nervous system disease
5. Known active plasma cell neoplasm, prolymphocytic leukemia, T-cell lymphoma, Burkitt lymphoma, acquired immunodeficiency syndrome (AIDS)-related B-cell lymphoma, Castleman disease, post-transplant lymphoproliferative disorders, hairy cell leukemia, germinal center B-cell (GCB), DLBCL, EBV+ DLBCL NOS, primary DLBCL of the central nervous system (CNS), primary cutaneous DLBCL - leg type, DLBCL associated with chronic inflammation, primary mediastinal (thymic) large B-cell lymphoma, intravascular large B-cell lymphoma, ALK+ large B-cell lymphoma, primary effusion lymphoma, high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements, high-grade B-cell lymphoma - NOS, B-cell lymphoma unclassifiable with features intermediate between DLBCL and classical Hodgkin lymphoma, or history of or currently suspected transformation of an indolent lymphoma to an aggressive histology (except for participants with Richter Transformation to DLBCL are eligible for Part 1a, 1c, or Phase 2 and participants with history of follicular lymphoma transforming to non-GCB DLBCL who are eligible for Part 1a, 1c, or Phase 2).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Participants with Adverse Events (AEs) | From the first dose of BGB-16673 until 30 days after the last dose of the study drug or before the initiation of a new anticancer therapy, whichever occurs first (Up to 47 weeks)
  Number of participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) including results from laboratory assessments, electrocardiograms (ECGs), and physical examinations, and that meet protocol-defined dose-limiting toxicities (DLTs); as graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.
Phase 1: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BGB-16673 | Approximately 28 days
  MTD is defined as the highest evaluated dose with an estimated toxicity rate closest to the target, while MAD is the highest dose given if MTD is not reached.
Phase 1: Recommended dose(s) for Expansion (RDFE) of BGB-16673 | Approximately 3 years
  RDFE of BGB-16673 alone will be determined based upon the MTD or MAD.
Phase 2: Overall response rate (ORR) | approximately 3 years
  Defined as the percentage of participants achieving a best overall response of partial response (PR) or better, assessed by the Independent Review Committee for participants with R/R CLL/SLL and R/R WM (in participants with WM, this is also referred to as major response rate) and by the investigator for other cohorts (R/R MCL, R/R MZL, R/R FL, R/R non-GCB DLBCL, R/R Richter's transformation to DLBCL), evaluated using the Lugano criteria for NHL and SLL, International Workshop of Chronic Lymphocytic Leukemia (iwCLL) criteria for CLL, and the 11th International Workshop on Waldenstrom's Macroglobulinemia (IWWM-11) criteria for WM.

SECONDARY OUTCOMES:
Single dose and steady-state maximum observed plasma concentration (Cmax) of BGB-16673 | Week 1 Day 1 pre-dose; 2, 4, 6, 8, 24, 48, and 72 hours post-dose; Week 5 Day 1 pre-dose; and 2, 4, 6, 8 post-dose; Week 9 Day 1 pre-dose.
Single dose and steady-state minimum observed plasma concentration (Cmin) of BGB-16673 | Week 1 Day 1 pre-dose; 2, 4, 6, 8, 24, 48, and 72 hours post-dose; Week 5 Day 1 pre-dose; and 2, 4, 6, 8 post-dose; Week 9 Day 1 pre-dose.
Single dose and steady-state time to reach Cmax (tmax) of BGB-16673 | Week 1 Day 1 pre-dose; 2, 4, 6, 8, 24, 48, and 72 hours post-dose; Week 5 Day 1 pre-dose; and 2, 4, 6, 8 post-dose; Week 9 Day 1 pre-dose.
Single dose and steady-state time to reach half of Cmax (T1/2) of BGB-16673 | Week 1 Day 1 pre-dose; 2, 4, 6, 8, 24, 48, and 72 hours post-dose; Week 5 Day 1 pre-dose; and 2, 4, 6, 8 post-dose; Week 9 Day 1 pre-dose.
Single dose and steady-state area under the plasma concentration-time curve (AUC) of BGB-16673 | Week 1 Day 1 pre-dose; 2, 4, 6, 8, 24, 48, and 72 hours post-dose; Week 5 Day 1 pre-dose; and 2, 4, 6, 8 post-dose; Week 9 Day 1 pre-dose.
Single dose and steady-state apparent total clearance of drug from plasma after oral administration (CL/F) of BGB-16673 | Week 1 Day 1 pre-dose; 2, 4, 6, 8, 24, 48, and 72 hours post-dose; Week 5 Day 1 pre-dose; and 2, 4, 6, 8 post-dose; Week 9 Day 1 pre-dose.
Single dose and steady-state apparent volume of distribution (Vz/F) of BGB-16673 | Week 1 Day 1 pre-dose; 2, 4, 6, 8, 24, 48, and 72 hours post-dose; Week 5 Day 1 pre-dose; and 2, 4, 6, 8 post-dose; Week 9 Day 1 pre-dose.
Single dose and steady-state accumulation ratios of BGB-16673 | Week 1 Day 1 pre-dose; 2, 4, 6, 8, 24, 48, and 72 hours post-dose; Week 5 Day 1 pre-dose; and 2, 4, 6, 8 post-dose; Week 9 Day 1 pre-dose.
Bruton's tyrosine kinase (BTK) protein degradation in peripheral blood after BGB-16673 monotherapy | Week 1 Day 1 pre-dose; 8, 24, 48, and 72 hours post-dose; Week 5 Day 1 pre-dose and 8 hours post-dose; Week 9 Day 1 pre-dose.
Phase 1: Overall response rate (ORR) | approximately 3 years
  Defined as the percentage of participants whose best overall response is partial response or better, as assessed by the investigator and evaluated according to the following criteria: the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria for R/R CLL, the International Workshop on Waldenström's Macroglobulinemia (IWWM-11) criteria for R/R WM (in participants with WM, this is also referred to as major response rate), and the Lugano criteria for R/R NHL.
Phase 1: Response Rate in Participants with R/R CLL/SLL | approximately 3 years
  Defined as the percentage of participants with R/R CLL/SLL whose best overall response is better than stable disease, as determined by investigators.
Phase 1: Overall Response Rate in Participants with R/R WM | approximately 3 years
  Defined as the percentage of participants with R/R WM who have a response rate of minor response or better.
Phase 1: Number of Participants with AEs in part 1e (Japan-only cohort ) | From the first dose of BGB-16673 in Part 1e until 30 days after the last dose of the study drug or before the initiation of a new anticancer therapy, whichever occurs first (approximately 3 years)
  Number of Japanese participants in Part 1e with TEAEs and SAEs, including results from laboratory assessments, ECGs, and physical examinations, that meet protocol-defined DLTs, graded according to the NCI-CTCAE v5.0.
Phase 2: Recommended Phase 2 Dose (RP2D) | approximately 3 years
  The Recommended Phase 2 Dose (RP2D) is determined by the sponsor based on the Safety Monitoring Committee's recommendations, taking into account the overall clinical safety, efficacy, pharmacokinetic (PK), and pharmacodynamic data.
Phase 2: Number of Participants with AEs | From the first dose of BGB-16673 in Phase 2 until 30 days after the last dose of the study drug or before the initiation of a new anticancer therapy, whichever occurs first (approximately 3 years)
  Number of participants with TEAEs and SAEs, including results from laboratory assessments, ECGs, and physical examinations, graded according to the NCI-CTCAE v5.0.
Phase 2: ORR in Participants with CLL/SLL assessed by investigators | approximately 3 years
  Defined as the percentage of participants with CLL/SLL with a best overall response of PR or better, as determined by investigators.
Phase 2: Major Response Rate for Participants with WM assessed by investigator | approximately 3 years
  Defined as the percentage of participants with WM whose best overall response is PR or better, as determined by investigators using the IWWM-11 criteria.
Phase 2: Overall Response Rate for Participants with WM assessed by investigator and IRC | approximately 3 years
  Defined as the percentage of participants who achieve at least a minor response (MR) or a more favorable outcome, as assessed by investigators for participants with R/R WM.
Phase 2: Rate of Very Good Partial Response (VGPR) or Better in Participants with WM Assessed by Investigator and IRC | approximately 3 years
  Defined as the percentage of participants with R/R WM with best response of VGPR or better as determined by IRC and investigator.
Phase 2: Response Rate in Participants with R/R CLL/SLL Assessed by Investigator and IRC | approximately 3 years
  Defined as the percentage of participants with R/R CLL/SLL whose best overall response is better than stable disease, as determined by IRC and investigator.
Phase 2: Duration of Response (DOR) | approximately 3 years
  DOR is defined as the time from the date that response criteria are first met to the date that progressive disease is documented or death, whichever comes first as assessed by the investigator and the IRC.
Phase 2: Time to Overall Response (TTOR) | approximately 3 years
  TTOR is defined as the time from study treatment start to date of the earliest qualifying response (partial response or better), as assessed by IRC and the investigator
Phase 2: Time to Major Response (TTMR) in Participants with WM | approximately 3 years
  Defined as the time from the date of treatment initiation to the date of first response of PR or better in participants with R/R WM.
Phase 2: Time to Response in Participants with R/R CLL/SLL Assessed by Investigator and IRC | approximately 3 years
  Defined as the time to first response based on best overall response of better than stable disease, per IRC and investigator.
Phase 2: Time to Response in Participants with WM Assessed by Investigator and IRC | approximately 3 years
  Defined as the time to first response based on best overall response of minor response or better, per IRC and investigator.
Phase 2: Time to Next Treatment (TTNT) | approximately 3 years
  Defined as the time from the treatment start date to the initiation of subsequent anticancer therapy.
Phase 2: Progression- Free Survival (PFS) | approximately 3 years
  PFS is defined as the time from first dose until first documentation of progression or death, whichever comes first, as assessed by IRC for R/R CLL/SLL and R/R WM and by the investigator for all participants.
Phase 2: Overall Survival (OS) | approximately 3 years
  OS is defined as the time from first study drug administration to the date of death due to any cause
Phase 2: Functional Assessment of Cancer Therapy-Leukemia (FACT-Leu) questionaire | Baseline and day 1 of Weeks 5, 13, 25, and 37
  Mean change from baseline in the 'physical well-being' and 'functional well-being' subscales of the FACT-Leu for participants with R/R CLL/SLL. FACT-Leu is a 44-item PRO questionnaire with five subscales used to measure health-related quality of life (HRQoL) in leukemia patients.
Phase 2: National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Lymphoma Cancer Symptom Index - 18 (NFLymSI-18) | Baseline and day 1 of Weeks 5, 13, 25, and 37
  Mean change from baseline in the NFlymSI-18 subscales of disease-related symptoms (DRSP) and 'treatment side effects' for participants with R/R MCL and participants with R/R WM. The NFlymSI-18 is an 18-item patient-reported outcome (PRO) tool specifically designed to assess symptoms and treatment impacts in patients with non-Hodgkin lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (113):
- United States (31):
  - University of Alabama At Birmingham Hospital, Birmingham, Alabama
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Honor Health Research Institute, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of California San Diego (Ucsd) Moores Cancer Center, La Jolla, California
  - Stanford Medicine, Palo Alto, California
  - UCLA Santa Monica Cancer Care, Santa Monica, California
  - Uchealth North, Fort Collins, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Tampa General Hospital Cancer Institute, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Midwestern Regional Medical Center, Zion, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton Cancer Institute Pavilion, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - American Oncology Partners of Maryland Pa, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College Newyork Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center Mskcc, New York, New York
  - Tennesse Oncology Chattanooga Downtown, Chattanooga, Tennessee
  - Tennessee Oncology, Pllc Nashville, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (9):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
  - Perth Blood Institute, West Perth, Western Australia
- Brazil (9):
  - Hospital Sirio Libanes Brasilia, Brasília
  - Hospital Erasto Gaertner, Curitiba
  - Centro Gaucho Integrado de Oncologia Hospital Mae de Deus, Porto Alegre
  - Real E Benemerita Associacao Portuguesa de Sao Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Hospital Nove de Julho Dasa, São Paulo
  - Instituto Dor de Pesquisa E Ensino Sao Paulo, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
  - Hospital Santa Rita de Cassia Afecc, Vitória
- Canada (5):
  - Arthur Je Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency the Vancouver Centre, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Chu de Quebec Universite Laval, Hopital de Lenfant Jesus, Centre Integre de Cancerologie (Cic), Québec
- China (4):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Guangxi Medical University Cancer Hospital Wuxiang Branch, Nanning, Guangxi
  - Yichang Central Peoples Hospitaljiangnan Branch, Yichang, Hubei
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciencestuanbo Branch, Tianjin, Tianjin Municipality
- France (9):
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Hopital Estaing, Clermontferrand
  - Chu Henri Mondor, Créteil
  - Hopital Claude Huriez Chu Lille, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Chu Montpellier Hopital Saint Eloi, Montpellier
  - Hopital de La Pitie Salpetriere, Paris
  - Centre Henri Becquerel, Rouen
- Arensia Exploratory Medicine Llc, Tbilisi, Georgia
- Germany (7):
  - Uniklinik Koeln (Aoer), Cologne
  - Universitatsklinikum Carl Gustav Carus An Der Technischen Universitat Dresden, Dresden
  - Universitares Krebszentrum Leipzig, Leipzig
  - Universitaetsklinikum Schleswig Holstein Campus Luebeck, Lübeck
  - Klinikum Johannes Gutenberg Universitaet Mainz, Mainz
  - Klinikum Grosshadern Ludwig Maximilians Universitat Munchen, München
  - Universitaetsklinikum Ulm, Ulm
- Italy (6):
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Ospedale San Raffaele, Milan
  - Istituto Europeo Di Oncologia, Milan
  - Niguarda Cancer Center Division of Hematology, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Centroricerche Cliniche Di Verona Srl, Verona
- Japan (5):
  - Aichi Cancer Center Hospital Clinical Oncology, Nagoya, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Cancer Institute Hospital of Jfcr, Kotoku, Tokyo
  - Yokohama Municipal Citizens Hospital, Yokohama
- The Institute of Oncology, Arensia Exploratory Medicine, Chisinau, Moldova
- South Korea (7):
  - Inje University Busan Paik Hospital, BusanjinGu, Busan Gwang'yeogsi
  - Pusan National University Hospital, Seogu, Busan Gwang'yeogsi
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi
- Spain (7):
  - Hospital Universitario Vall Dhebron, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Md Anderson Cancer Center Madrid Spain, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (2):
  - Sahlgrenska University Hospital Hematology, Gothenburg
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Turkey (Türkiye) (4):
  - Dokuz Eylul University, Balçova
  - Erciyes University, Kayseri
  - Sakarya Training and Research Hospital, Sakarya
  - Ondokuz Mayis University, Samsun
- United Kingdom (6):
  - Edinburgh Cancer Centre, Edinburgh
  - Churchill Hospital Oxford University Hospital Nhs Trust, Headington
  - St Jamess University Hospital, Leeds
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospitals Nhs Trust, Nottingham
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/